CLINICAL TRIAL: NCT03230929
Title: The Effect of EMG Activity on Anesthetic Depth Monitoring : Comparison Between Phase Lag Entropy and BIS
Brief Title: The Effect of Electromyogram (EMG) Activity on Anesthetic Depth Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Tae-Kyun Kim, Associate Professor, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: L-2017-165
Record Dates: First submitted 2017-07-16; First posted 2017-07-27 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: General Anesthetic Drug Overdose
Keywords: EMG, BIS, phase lag entropy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIS-PLE (Experimental): Anesthesiologist attaches the sensors of BIS and PLEM 100 on the forehead of the patient, and monitor the monitor and record the values of BIS, PLEM 100, and neuromuscular monitoring.
  Interventions: Device: BIS-PLE

INTERVENTIONS:
Device: BIS-PLE — Anesthesiologist attaches the sensors of BIS and PLEM 100 on the forehead of the patient, and adheres the neuromuscular monitoring device on the medial side of the wrist and the ipsilateral thumb to continuously monitor the state of consciousness and muscle relaxation before, during and after surgery. Reversal of muscle relaxant could be performed by intravenous injection of sugammadex 4 mg/ kg in the case of deep neuromuscular relaxation, and 2 mg / kg in the case of shallow muscle relaxation degree under neuromuscular monitoring. After then, they monitor and record the values of BIS, PLEM 100, and neuromuscular monitoring in 1 minute increments for 5 minutes.

SUMMARY:
Currently, a lot of equipments based on Bispectral index (BIS) is used clinically in order to measure the depth of anesthesia. Although BIS is used for the measurement of the presence of consciousness or degree of sedation during general anesthesia, it could be influenced by factors that affect or interfere with the activity of EEG because it is a numerical value which is measured by analyzing EEG. The BIS electrode for EEG analysis should be attached to the patient's forehead and the EEG signal is 0.5 - 30 Hz, the EMG signal is 30 - 300 Hz, and the BIS analyzes the 0 - 47 Hz signal. Therefore, 30 -47 Hz EMG signal may influence the BIS value and the BIS value may differ from the actual. In patients with complete muscle relaxation, the change in BIS varies in proportion to the concentration of anesthetic, but in a state with less muscle relaxation or arousal period of anesthesia when recovery of muscle relaxation occurs, BIS value may not accurately reflects the change in the depth of anesthesia. Although there is a study on the influence of the degree of muscle relaxation on BIS value, there is no study on whether phase lag entropy (PLE) measuring anesthesia depth based on different mechanism from BIS is affected by status of muscle relaxation. After measuring BIS and PLE at the same time, I will compare both of them and investigate the reliability of the measurement of the depth of anesthesia of PLE and how electromyogram activity affects PLE.

DETAILED DESCRIPTION:
Intravenous administration of 2% propofol and remifentanil would be done for total intravenous anesthesia. After intravenous injection of rocuronium 0.6 mg/ kg for muscle relaxation, endotracheal intubation would be performed. Then, anesthesiologist attaches the sensors of BIS and PLEM 100 on the forehead of the patient, and adheres the neuromuscular monitoring device on the medial side of the wrist and the ipsilateral thumb to continuously monitor the state of consciousness and muscle relaxation before, during and after surgery. Before the end of surgery, the degree of neuromuscular relaxation should be within deep block (TOF count <2) and the concentration of 2% propofol should be adjusted for maintaining BIS between 50 and 60. Reversal of muscle relaxant could be performed by intravenous injection of sugammadex 4 mg/ kg in the case of deep neuromuscular relaxation, and 2 mg / kg in the case of shallow muscle relaxation degree under neuromuscular monitoring. After then, monitor and record the values of BIS, phase lag entropy monitor (PLEM) 100, and neuromuscular monitoring in 1 minute increments for 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* The patient who is scheduled for operation requiring general anesthesia and whose American Society of Anesthesiologists (ASA) status is I or II.

Exclusion Criteria:

* Who has neuromuscular disease
* Who takes medicines related neurologic system

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
The difference of phase lag entropy between before and after neuromuscular recovery | 24 hours
  PLEM 100 is 4-channel electroencephalogram (EEG) monitor and it records electric activity signals of the brain generated from the human body. The anesthesiologist administers sugammadex intravenously at the end of the surgery, and then monitors and records the values of BIS, PLEM 100, and neuromuscular monitoring in 1 minute increments for 5 minutes until neuromuscular recovery is completed.

SECONDARY OUTCOMES:
The difference between BIS and phase lag entropy during general anesthesia | 24 hours
  BIS uses the frequency, amplitude, phase angle of electroencephalogram, and measures the coherence. Finally, it is closely related to the level of sedation and consciousness by the anesthetic agent. PLEM 100 is 4-channel electroencephalogram monitor and it records electric activity signals of the brain generated from the human body. The anesthesiologist continuously monitor the state of consciousness and muscle relaxation from entrance of the patient to the complete recovery of muscle relaxation.

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Kyun Kim, PhD., Principal Investigator — Pusan National University Yangsan Hospital, Geumo-ro 20, Mulgeum-eup, Yangsan, 50612
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT03230929/Prot_003.pdf
  • Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT03230929/SAP_004.pdf
  • Informed Consent Form (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT03230929/ICF_005.pdf